CLINICAL TRIAL: NCT05525117
Title: Evaluating the Effectiveness of an Online Self-management Intervention for Type 2 Diabetes Mellitus (Covivio): Randomized Controlled Trial
Brief Title: Effectiveness of an Online Self-management Intervention for Type 2 Diabetes Mellitus
Acronym: OnSeT-2D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants could be recruited.
Sponsor: Gaia AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: covivio trial 2022
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; covivio; diabetes self-management; digital health application
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with two arms: (i) online intervention in addition to treatment-as-usual versus (ii) treatment-as-usual
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online intervention in addition to treatment-as-usual (Experimental): online intervention: covivio in addition to treatment as usual
  Interventions: Behavioral: covivio (additional to treatment as usual)
- treatment-as-usual (Other): Other: treatment as usual
  Interventions: Other: treatment as usual

INTERVENTIONS:
Behavioral: covivio (additional to treatment as usual) — Covivio is a dialogue-based online psychological intervention for patients with type 2 diabetes. This intervention includes elements that address disease literacy, physical activity and exercise, dieting and nutritional principles, coping with depression, etc. Content is adapted to users needs using interactive dialogues, illustrations and audio files. Participants may also continue with their usual treatment.
  Arms: online intervention in addition to treatment-as-usual
Other: treatment as usual — Participants may continue with any treatment that they require (treatment as usual)
  Arms: treatment-as-usual

SUMMARY:
This trial was designed to evaluate the effectiveness of the dialogue-based online intervention covivio, which was designed to improve diabetes self-management in patients with type 2 diabetes.

The study aims to test the hypothesis that covivio has a greater positive impact on glycemic control than treatment as usual. Patients with type 2 diabetes mellitus will be randomized and allocated to either an intervention group, receiving covivio in addition to treatment as usual, or a control group, which receives only treatment as usual. The primary endpoint is the HbA1c value six month after baseline.

DETAILED DESCRIPTION:
The aim of this clinical trial is to investigate the effectiveness of the self-guided digital therapeutic covivio in 268 patients with type 2 diabetes mellitus (T2DM). Patients will be randomized and allocated in a 1:1 ratio to either an intervention group, in which they will receive access to covivio in addition to treatment as usual (TAU, n = 134), or to a control group, in which they will receive only TAU (n = 134).

The primary endpoint of this trial will be the between-groups difference of the HbA1c in the intervention and control group at six months adjusted for the baseline HbA1c. In order to show the course of change over time, two timepoints for assessment of effects are planned at four (T1) and six months (T2) after the baseline assessment (T0). The primary endpoint will be the HbA1c at six months post-allocation. Secondary endpoints will be depression, diabetes self-management (DSM), BMI, and quality of life. Figure 1 (section 6.1) summarizes the design of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of T2DM (submission of a medical certificate attesting to the presence of at least one of the following ICD-10-GM diagnoses of T2DM: E11.20, E11.30, E11.40, E11.50, E11.60, E11.72, E11.74, E11.80, E11.90)
* HbA1c value ≥ 7.0% (53 mmol/mol)
* BMI ≥ 23 kg/m2
* Consent to participate
* Sufficient knowledge of the German language

Exclusion Criteria:

* diagnosis of type 1 diabetes mellitus (T1DM)
* change in medication, frequency of use or dosage (planned within 4 weeks before T0 or during the study period)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  The primary objective of this study is to determine whether the online intervention covivio will reduce HbA1c values in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Depressive symptoms | 6 months
  assessed with the total score of the Patient Health Questionnaire (PHQ-9)
Diabetes Self-management | 6 months
  assessed with the total mean score of the Diabetes Self-management questionnaire (DSMQ)
Body Mass Index | 6 months
  calculated from measurement data of patient's height in meter and weight in kilogram
Health-Related Quality of Life | 6 months
  assessed with the total score of the Assessment of Quality of Life (AQoL-8D)
Proportion of patients achieving a reduction in HbA1c | 6 months
  A reduction of HbA1c values by at least 0.3% from baseline to T2 will be considered a significant clinical improvement in glycemic control

OTHER OUTCOMES:
Waist circumference | 6 months
  measured at the midpoint between the lower rib and iliac crest in centimeters
systolic blood pressure | 6 months
  measured with a calibrated sphygmomanometer while the subject is sitting

CONTACTS AND LOCATIONS:
Overall Officials: Gitta Jacob, PD PhD, Principal Investigator — Gaia AG
Locations (1):
- GAIA, Hamburg, Germany